CLINICAL TRIAL: NCT04697576
Title: Intralesional Influenza Vaccine for Patients With Melanoma
Brief Title: Intralesional Influenza Vaccine for the Treatment of Stage I-IV Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Carlo Contreras (Other)
Responsible Party: Sponsor-Investigator, Carlo Contreras, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20221; NCI-2020-13282 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Clinical Stage I Cutaneous Melanoma AJCC v8; Clinical Stage IA Cutaneous Melanoma AJCC v8; Clinical Stage IB Cutaneous Melanoma AJCC v8; Clinical Stage II Cutaneous Melanoma AJCC v8; Clinical Stage IIA Cutaneous Melanoma AJCC v8; Clinical Stage IIB Cutaneous Melanoma AJCC v8; Clinical Stage IIC Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; pembrolizumab; Influenza Vaccines; relatlimab; Opdualag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (resectable Stage I-III melanoma) (Experimental): Patients receive an influenza vaccine IM on day 0 and intratumorally on days 2 and 14 in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery on day 28.
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine; Procedure: Resection
- Cohort II (unresectable Stage IV) (Experimental): Patients receive an influenza vaccine IM on day 0 and intratumorally on days 2, 14, 28, 42, 56, 70, 84, and 98 in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care (single- or dual-agent) ipilimumab, nivolumab, relatlimab, or pembrolizumab.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Biological: Pembrolizumab; Biological: Quadrivalent Inactivated Influenza Vaccine; Biological: Nivolumab + Relatlimab

INTERVENTIONS:
Biological: Ipilimumab — immune checkpoint inhibitor
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Cohort II (unresectable Stage IV)
Biological: Nivolumab — immune checkpoint inhibitor
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Cohort II (unresectable Stage IV)
Biological: Pembrolizumab — immune checkpoint inhibitor
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Cohort II (unresectable Stage IV)
Biological: Quadrivalent Inactivated Influenza Vaccine — Given IM and intratumorally. For this protocol the U.S. F.D.A recently approved the use of recently expired influenza vaccine (only until new seasonal vaccine is available anticipated Sept 1). Use of expired vaccine will not exceed 4 months past June 30th expiry date (October 30th).
  Other Names: Fluzone Quadrivalent; Fluzone Quadrivalent Influenza Vaccine; QIV; Quadrivalent Influenza Vaccine
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
  Arms: Cohort I (resectable Stage I-III melanoma)
Biological: Nivolumab + Relatlimab — immune checkpoint inhibitor
  Other Names: Opdualag
  Arms: Cohort II (unresectable Stage IV)

SUMMARY:
This phase I trial investigates the effects of influenza vaccine in treating patients with stage I-IV melanoma. While intramuscular administration of influenza vaccine provides immunization against the influenza virus, giving influenza vaccine directly into the tumor (intralesional) may decrease the size of the injected melanoma tumor, or the extent of the melanoma within the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability and determine the maximum tolerated dose of intralesional (quadrivalent inactivated influenza vaccine (unadjuvanted influenza vaccine) for patients with a) resectable melanoma as monotherapy, and b) metastatic melanoma, concurrent with standard of care (single- or dual-agent) checkpoint inhibition.

SECONDARY OBJECTIVES:

I. To evaluate tumor dimensions of injected (Cohorts #1-2) and non-injected lesions (Cohort #2 only), by caliper or ultrasound measurement. (Clinical endpoint) II. To determine time to disease progression (local or distant). (Clinical endpoint) III. To evaluate immunohistochemistry density, cells/mm^2: CD4, CD8, PD-L1, PD1, CD56, CD20, CD45RO, FOXP3. (Tumor-based endpoint) IV. To evaluate granzyme B H-score. (Tumor-based endpoint) V. To evaluate NanoString Pan Cancer Immune Profiling Panel. (Tumor-based endpoint) VI. To evaluate tumor-infiltrating lymphocytes: not identified, present (non-brisk), present (brisk), cannot be determined. (Tumor-based endpoint) VII. To evaluate degree of tumor regression (percent). (Tumor-based endpoint) VIII. To evaluate changes in micro ribonucleic acid (microRNA) expression. (Tumor-based endpoint) IX. To evaluate of flow cytometry for T-cell subset evaluation and changes in circulating microRNA. (Blood draw endpoint)

EXPLORATORY OBJECTIVE:

I. To evaluate the evidence of immunologic activation in blood and tissue specimens.

OUTLINE: This is dose-escalation study. Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive quadrivalent inactivated influenza vaccine intramuscularly (IM) on day 0 and intratumorally on days 2 and 14 in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery on day 28.

COHORT II: Patients receive quadrivalent inactivated influenza vaccine IM on day 0 and intratumorally on days 2, 14, 28, 42, 56, 70, 84, and 98 in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care ipilimumab, nivolumab, pembrolizumab, or Opdualag.

After completion of study treatment, patients are followed up for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* 18 to 99 years of age
* Histologically confirmed cutaneous melanoma by historical pathology report review, clinical Stage I-III (Cohort #1), or Stage IV (Cohort #2) cutaneous melanoma
* At least one, biopsy-proven, palpable melanoma tumor deposit suitable for intralesional injection measuring ≥ 1 cm by digital caliper (with digital photography documentation) or ultrasound (with ultrasound image documentation)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Absolute neutrophil count (ANC) >= 1.5 x 10^3/mm^3 (drawn at or not more than 30 days prior to the screening visit)
* Hemoglobin (Hgb) >= 9 g/dL (drawn at or not more than 30 days prior to the screening visit)
* Platelet count >= 100 x 10^3/mm^3 (drawn at or not more than 30 days prior to the screening visit)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) or =< 5 x ULN in patients with liver metastases (Cohort 2 only) (drawn at or not more than 30 days prior to the screening visit)
* Prothrombin time =< 1.5 x ULN (drawn at or not more than 30 days prior to the screening visit)
* Total bilirubin =< 1.5 x ULN (unconjugated bilirubin of < 3 x ULN for patients with known Gilbert syndrome) (drawn at or not more than 30 days prior to the screening visit)
* Creatinine clearance of >= 50 ml/min by Cockcroft-Gault equation (drawn at or not more than 30 days prior to the screening visit)
* Women of childbearing potential (WOCBP) must agree to use effective contraceptive methods from screening until at least:

  * Cohort 1: 14 days after the surgical resection for subjects in Cohort 1
  * Cohort 2:

    * Nivolumab: 5 months after the last dose of either nivolumab or intralesional Flucelvax, whichever is later
    * Pembrolizumab: 4 months after the last dose of either pembrolizumab or intralesional Flucelvax, whichever is later
    * Ipilimumab: 3 months after the last dose of either ipilimumab or intralesional Flucelvax, whichever is later
    * Relatlimab + nivolumab (marketed under the trade name Opdualag): 5 months after the last dose of either Opdualag or intralesional Flucelvax, whichever is later.
    * Combination ipilimumab with other checkpoint inhibitor: Whichever is later:

      * 3 months after the last dose of either ipilimumab or intralesional Flucelvax
      * Above-bulleted recommendation for nivolumab or pembrolizumab
* Non-childbearing potential is defined as a woman who meets either of the following criteria: a) postmenopausal state defined as no menses for 12 months without an alternative medical cause, or b) documented hysterectomy, bilateral tubal ligation, or bilateral oophorectomy
* Effective contraception methods are defined as one of the following:

  * True abstinence, defined as refraining from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject
  * Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception
  * Condoms and spermicide
  * Diaphragm and spermicide
  * Oral or implanted hormonal contraceptive
  * An intra-uterine device
* WOCBP must have a negative pregnancy test (serum or urine)

Exclusion Criteria:

* Known allergy or intolerance to influenza vaccination
* Subjects with condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone/equivalent) or other immunosuppressive medications within 14 days of study drug administration
* Active, known or suspected autoimmune disease
* Active brain metastasis or leptomeningeal metastasis
* Diagnostic biopsy of ocular or mucosal melanoma
* Any melanoma therapy within 6 months of enrollment; though prior surgical resection is permitted
* Incarcerated patients
* Patients known to be HIV positive are eligible if they meet the following criteria within 30 days prior to randomization: stable and adequate CD4 counts (≥ 350 mm^3), and serum HIV viral load of < 25,000 IU/ml. Patients may be on or off anti-viral therapy so long as they meet the CD4 count criteria
* Pregnant or lactating patients
* Patients incapable of independently providing consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 1 year after the last intra-tumoral dose
  Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. All patients who have received at least one dose of the therapeutic agents will be evaluable for toxicity and tolerability.
Maximum tolerated dose (MTD) in Cohorts #1 and #2 | Up to 98 days
  Will employ the Bayesian optimal interval design to find the MTD.

SECONDARY OUTCOMES:
Tumor dimensions of injected (Cohorts #1) | Up to 1 year after the last intra-tumoral dose
  Will be assessed by caliper or ultrasound measurement. Tumor dimensions will be summarized using descriptive statistics (i.e. mean with standard deviations, or median with range).
Tumor dimensions of non-injected lesions (Cohort #2) | Up to 1 year after the last intra-tumoral dose
  Will be assessed by caliper or ultrasound measurement. Tumor dimensions will be summarized using descriptive statistics (i.e. mean with standard deviations, or median with range).
Time to disease progression (local or distant) | From the start of treatment until the documentation of local or distant disease progression, assessed up to 1 year
  Time to disease progression will be analyzed using Kaplan-Meier method, resulting in median survival times with 95% confidence interval, assuming sufficient events have occurred.
Biomarker analysis | Up to 1 year after the last intra-tumoral dose
  Will analyze immunohistochemistry density, cells/mm^2 of CD4, CD8, PD-L1, PD1, CD56, CD20, CD45RO, FOXP3. Summary statistics will be used.
Granzyme B H-score | Up to 1 year after the last intra-tumoral dose
  Summary statistics will be used.
NanoString Pan Cancer Immune Profiling Panel | Up to 1 year after the last intra-tumoral dose
  Summary statistics will be used.
Tumor-infiltrating lymphocytes analysis | Up to 1 year after the last intra-tumoral dose
  Will analyze tumor-infiltrating lymphocytes: not identified, present (non-brisk), present (brisk), cannot be determined. Summary statistics will be used.
Degree of tumor regression (percent) | Up to 1 year after the last intra-tumoral dose
  Summary statistics will be used.
Changes in micro ribonucleic acid (RNA) expression | Baseline up to 1 year after the last intra-tumoral dose
  Summary statistics will be used.
T-cell subset evaluation and changes in circulating microRNA | Up to 1 year after the last intra-tumoral dose
  Summary statistics will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo M Contreras, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu